CLINICAL TRIAL: NCT02885545
Title: The Strategy to Prevent Hemorrhage Associated With Anticoagulation in Renal Disease Management (STOP HARM) Trial
Acronym: STOP-HARM
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Failure to recruit any participants in more than one year of recruiting.
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STOP HARM
Record Dates: First submitted 2016-06-24; First posted 2016-08-31 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: Chronic Kidney Disease; Acute Bleeding; Cerebrovascular Stroke
MeSH Terms: conditions — Renal Insufficiency, Chronic; Stroke | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Left atrial appendage occlusion (Experimental): Patients receiving the Watchman device will have it placed via a percutaneous trans-septal approach under transesophageal echocardiographic and fluoroscopic guidance. Patients will be anticoagulated for at least 45 days after the procedure.
  Interventions: Device: Watchman
- Continuation of prescribed anticoagulant (Active Comparator): Patients continuing medical therapy will continue to take their previously prescribed oral anticoagulation (vitamin K antagonist, apixiban or rivaroxaban) for the duration of the study unless a medical reason to alter therapy occurs.
  Interventions: Drug: Continued therapy with the prescribed oral anticoagulant

INTERVENTIONS:
Device: Watchman — If the patient is randomized to the Intervention Arm of the study the Watchman device will be implanted into the left atrial appendage of the heart
  Arms: Left atrial appendage occlusion
Drug: Continued therapy with the prescribed oral anticoagulant — If the patient is randomized to the control arm of the study, they will continue taking the oral anticoagulant that has been prescribed (vitamin K antagonist, Apixiban 2.5mg bid or Rivaroxaban 15mg od)
  Other Names: Standard of care
  Arms: Continuation of prescribed anticoagulant

SUMMARY:
Patients with severe chronic kidney disease (CKD) who develop atrial fibrillation are at high risk for stroke. The use of blood thinking medication in dialysis patients is controversial and warfarin carries a serious risk for major bleeding.

The Watchman device may be an ideal therapy for this population as after implantation it allows for the discontinuation of blood thinners, thereby reducing the risk of bleeding.

DETAILED DESCRIPTION:
An estimated 25 million North American's have chronic kidney disease (CKD) including 600,000 that require dialysis for end-stage renal disease.The importance of CKD is underscored by the poor survival, frequent hospitalizations and impaired health related quality of life of patients with CKD.

Stroke is an important cause of morbidity, mortality and suffering for patients with CKD. Stroke is approximately 5 to 10 times more common in patients with advanced CKD compared to non-CKD patients. Atrial fibrillation (AF), the most important risk factor for stroke, occurs in up to 20.4% of patients with advanced CKD. Observational studies suggest anywhere from an approximate 56% relative risk reduction to a 2-fold increase in the risk of stroke with warfarin. Furthermore, the risk of bleeding in patients with advanced CKD is roughly 5-fold higher than patients without CKD. Although OAC may not prevent strokes in patients with advanced CKD, it still increases the risk of major bleeding by 1.4 fold.

New stroke prevention strategies in patients with CKD and AF are urgently needed. An effective strategy must reduce the risk of thromboembolic events while not increasing the risk of bleeding substantially. Left atrial appendage occlusion (LAAO) with devices such as the Watchman, represent a unique opportunity to accomplish effective stroke prevention while mitigating the risk of bleeding in this patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Severe chronic kidney disease: a. Receiving dialysis >90 days or b. Estimated glomerular filtration rate less than 30 ml/min/1.73m2 for >90 days as calculated by CKD-Epi
3. History of persistent, paroxysmal or permanent atrial fibrillation documented by ECG within 12 months of randomization
4. High risk of stroke: a. CHADS-VASC≥3 or, b. Prior ischemic stroke or TIA 2-24 months prior to randomization,
5. Currently receiving chronic oral anticoagulation (vitamin K antagonist, Apixaban 2.5 mg bid or Rivaroxaban 15mg od) for atrial fibrillation
6. Provides informed consent

Exclusion Criteria:

1. Short life expectancy: a. > 90 years old or, b. Positive "surprise" question (Physician not surprised if patient died in the next 12 months)
2. Stroke within the last 2 months
3. Contraindications to withdrawal of anticoagulation (e.g. mechanical valve, recurrent venous thromboembolism)
4. Contraindication to low-dose aspirin
5. Contraindication to placement of Watchman device: a. Thrombus formation in left atrial appendage b. Severe mitral or aortic valvular disease c. Left atrial appendage diameter too small or too large to accommodate the device d. Pericardial effusion >2 mm e. Cardiac tumor
6. Scheduled living related donor transplant

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-09 (Estimated); Primary Completion 2018-03-05 (Actual); Study Completion 2018-03-05 (Actual)

PRIMARY OUTCOMES:
Time from randomization to the first occurrence of major bleeding. | Approximately 5 years
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.

SECONDARY OUTCOMES:
Time from randomization to the first occurrence of ischemic stroke | Approximately 5 years
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Time from randomization to the first occurrence of either ischemic stroke or non-central nervous system arterial embolism | Approximately 5 years
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Time from randomization to the first occurrence of all-cause mortality | Approximately 5 years
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Time from randomization to the first occurrence of a life threatening bleed | Approximately 5 years
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Bleeding directly caused by implantation of Watchman Device | 30 days
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Device complications directly caused by implantation of Watchman Device | 30 days
  This evaluation will be based on a structured interview with the patient. In case of positive evaluation for the outcome more information will be obtained by hospital or physician.
Health related quality of life (EQ-5D-5L) | Approximately 5 years
  This evaluation will be based on a structured interview with the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Morillo, MD, Principal Investigator — Population Health Research Institute
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided